CLINICAL TRIAL: NCT01665768
Title: A Trial of Maintenance Rituximab With mTor Inhibition After High-dose Consolidative Therapy in CD20+, B-cell Lymphomas, Gray Zone Lymphoma, and Hodgkin's Lymphoma
Brief Title: Maintenance Rituximab With mTor Inhibition After High-dose Consolidative Therapy in Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1228; NA_00067315 (Other: JHMIRB)
Record Dates: First submitted 2012-07-27; First posted 2012-08-15 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: CD20+, B-cell Lymphomas; Mantle Cell Lymphoma; Non-Mantle Cell Low Grade B Cell Lymphomas (SLL/CLL); Transformed Lymphoma/DLBCL/PMBCL; Hodgkin's Disease; Gray Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Mantle-Cell; Hodgkin Disease | interventions — Everolimus; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus and Rituximab (Experimental): Everolimus daily for one year and IV rituximab four times during that year.
  Interventions: Drug: Everolimus; Biological: Rituximab

INTERVENTIONS:
Drug: Everolimus — The initial dose of everolimus will be 2.5mg orally daily for a total of one year to maintain a target trough concentration between 3-15 ng/mL.
  Other Names: RAD001
Biological: Rituximab — 375mg/m2 day +1 and then every 90 days for 1 year (a total of 4 infusions)
  Other Names: Rituxan

SUMMARY:
This research is being done to determine if combining an investigational drug called Everolimus with Rituximab can reduce the risk of your cancer from returning after high dose chemotherapy.

DETAILED DESCRIPTION:
Everolimus is a pill that interferes with lymphoma cell growth by blocking a cellular pathway important in causing cancer cells to grow, called mTor. Rituximab is an intravenous medication that specifically attacks a protein commonly found on lymphoma cells called CD20.

Rituximab is already widely used to treat multiple forms of lymphoma. Moreover, continuing rituximab after the completion of chemotherapy is already commonly used to help patients stay in remission longer. Everolimus has been shown in many types of relapsed lymphoma to decrease the size of lymph nodes by itself. Everolimus is approved by the Food and Drug Administration (FDA) for the treatment of advanced kidney cancer and subependymal giant cell astocytoma. It is not approved for use in lymphoma. The use of everolimus in this research study is investigational. The word "investigational" means that everolimus is not approved for marketing by the Food and Drug Administration (FDA). The FDA is allowing the use of everolimus in this study.

The combination of everolimus and rituximab for 1 year after high dose therapy is also new. We believe the combination of these medications right after your chemotherapy will be more effective in attacking your remaining cancer before they have time to re-grow.

The usual treatment of lymphoma after high-dose chemotherapy is observation. After your body has fully recovered from the effects of the chemotherapy, you will receive everolimus daily for one year and IV rituximab four times during that year.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years of age
* ECOG performance status ≤ 2
* INR ≤ 2
* Adequate renal and hepatic function defined as a serum creatinine <2.0mg/dL, total bilirubin <5mg/dL, and AST and ALT ˂ 2.5 ULN.
* Platelet count >75 x 109/L
* Hemoglobin >10mg/dL
* ANC >3.0x109/L
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L and fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* A willingness to use an accepted and effective method of birth control for sexually active women of childbearing potential during the study and for 8 weeks after the end of study drug treatment.
* Ability to sign informed consent

Exclusion Criteria:

Patient who have previously received an mTor inhibitor

* Patients who are pre-terminal or moribund
* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of Everolimus (including chemotherapy, radiation therapy, antibody based therapy, etc.)
* Uncontrolled diabetes mellitus as defined by HbA1c>8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary
* Chronic treatment with corticosteroids or other immunosuppressive agents. Topical or inhaled cortosteroids are allowed
* Patients who have received live attenuated vaccines within 1 week of start of Everolimus and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines;
* Patients who have a history of another primary solild malignancy, with the exceptions of: non-melanoma skin cancer, and carcinoma in situ of the cervix, uteri, or breast from which the patient has been disease free for ≥3 years;
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study;
* Patients with active bacterial or fungal infections requiring oral or intravenous antimicrobials are not eligible until resolution of the infection
* Female patients who are pregnant or breast feeding, or of reproductive potential whoe are not using effective birth control methods. Adequate contraception must be used throughout the trial and for 8 weeks after the last dose of study drug.
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Patients with known intolerance to rituximab
* Known history of HIV or Hepatitis C
* Active Hepatitis B as defined by seropositivity for hepatitis B surface antigen. Subjects with positive hepatitis B core antibody titers and normal liver transaminases are allowed provided that prophylaxis is administered per institutional guidelines. Please see Addendum 8 for the action to be taken for patients with positive baseline hepatitis B results.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Gladstone, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schoch LK, Asiama A, Zahurak M, Shanbhag S, Hurtt J, Sawyer K, Swinnen LJ, Wagner-Johnston N, Jones RJ, Ambinder RF, Gladstone DE. Pharmacokinetically-targeted dosed everolimus maintenance therapy in lymphoma patients. Cancer Chemother Pharmacol. 2018 Feb;81(2):347-354. doi: 10.1007/s00280-017-3499-y. Epub 2017 Dec 13. PMID 29234922

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 participants were screen failures.
Groups:
- Everolimus and Rituximab: Everolimus daily for one year and IV rituximab four times during that year.
  Everolimus: The initial dose of everolimus will be 2.5mg orally daily for a total of one year to maintain a target trough concentration between 3-15 ng/mL. Previously the study allowed for starting doses of 5mg and 10mg; the starting dose was reduced in subsequent amendments due to a high incidence of dose reductions. 2.5mg was the most frequent daily dose for all patients, and the entire population was analyzed as one arm.
  Rituximab: 375mg/m2 day +1 and then every 90 days for 1 year (a total of 4 infusions)
Period: Overall Study
Arm/Group | Everolimus and Rituximab
Started | 49
Completed | 26
Not Completed | 23
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 19
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus and Rituximab
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 12
Age, Continuous [Median (Full Range); unit: years] | 59 [36 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 43
  More than one race | 0
  Unknown or Not Reported | 3
Number of Prior Therapies [Count of Participants; unit: Participants]
  Two Prior Therapies | 30
  Three Prior Therapies | 18
  Four Prior Therapies | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety as Assessed by Avoidance of Grade 3-4 Adverse Events
Description: Number of participants who did not experience at least one grade 3-4 adverse event by CTCAE 4.0.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus and Rituximab
Number analyzed (Participants) | 49
Participants | 1

2. Secondary Outcome: Event Free Survival (EFS)
Description: Percentage of participants alive without disease progression. As defined by Cheson criteria, disease progression is a new lesion or >= 50% increase in the size of previously identified sites of disease. EFS was estimated using Kaplan-Meier survival analysis.
Time Frame: 2.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Everolimus and Rituximab
Number analyzed (Participants) | 49
percentage of participants | 58 [45 to 76]

3. Secondary Outcome: Percentage Change in the Frequency of Circulating Cancer Cells
Description: Percentage change in circulating cancer cells between baseline and each timepoint noted below.
Time Frame: Baseline, 1 year, 2 years and 3 years
Population: Data was not collected.
Arm/Group | Everolimus and Rituximab
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage Change in Cancer Cells When mTOR Kinase Inhibition is Applied
Description: Percentage change in cancer cells when mTOR inhibition is applied in the laboratory. Samples from participants will be evaluated at each timepoint noted below.
Time Frame: 1 year, 2 years, and 3 years
Population: Data was not collected.
Arm/Group | Everolimus and Rituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Adverse events were assessed every 2 weeks for the first 2 months, monthly for the remainder of the first year, every 90 days for the second year, and every 6 months for the third year. Per protocol, all adverse events were collected for the first 13 participants. Only grade 3-4 and all serious adverse events were collected for the remaining participants.
Arm/Group | Everolimus and Rituximab
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 13/49
Other Adverse Events (participants affected / at risk) | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus and Rituximab (N=49)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cellulitis (Infections and infestations) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Investigations) | 1 (1)
MRSA (Infections and infestations) | 1 (1)
Febrile neutropenia (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Retinal tear (Eye disorders) | 1 (1)
Zoster (Infections and infestations) | 1 (1)
Skin lesions (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus and Rituximab (N=49)
ALT increased (Investigations) | 4 (6)
Anemia (Investigations) | 5 (12)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Hyperglycemia (Investigations) | 10 (25)
Hypertriglyceridemia (Investigations) | 10 (17)
Insomnia (General disorders) | 3 (3)
Leukopenia (Investigations) | 31 (73)
Lymphopenia (Investigations) | 6 (15)
Mucositis (Skin and subcutaneous tissue disorders) | 4 (4)
Neuropathy (Nervous system disorders) | 4 (5)
Neutropenia (Investigations) | 29 (75)
Pain - throat (General disorders) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Thrombocytopenia (Investigations) | 8 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT01665768/Prot_SAP_000.pdf